CLINICAL TRIAL: NCT00726531
Title: Multi-centre Cluster Randomised Trial Comparing a Community Group Exercise Programme With Home Based Exercise With Usual Care for Over 65s in Primary Care
Brief Title: Promoting Physical Activity in the Over 65s
Acronym: ProAct65+
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Professor Steve Iliffe, University College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ProAct65+; UK HTA grant 06/36/04
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Falls
Keywords: Falls prevention; Exercise promotion; Older people
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OEP (Experimental): Home based exercise programme (OEP) This exercise programme consists of a 30 minute programme of leg muscle strengthening and balance retraining exercises progressing in difficulty to be performed at home at least three times per week, and a walking plan to be undertaken at least two times per week for 24 weeks. . Trained peer mentors will contact and visit the patients at their home to start the exercise programme with them and will follow-up with up to three more home visits / exercise sessions as the participants require
  Interventions: Behavioral: Otago Exercise Programme
- Fame (Experimental): Community based exercise programme (FaME) FaME includes and extends the OEP. It will comprise one hour PSI delivered group exercise class in a local community centre for a maximum of 15 participants, and two 30 minute home exercise sessions (based on the extended OEP) per week for 24 weeks. Participants will also be advised to walk at least twice per week for up to 30 minutes at a moderate pace.
  Interventions: Behavioral: Fame
- TAU (No Intervention): Treatment as usual
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Otago Exercise Programme — Home based exercise programme (OEP) This exercise programme consists of a 30 minute programme of leg muscle strengthening and balance retraining exercises progressing in difficulty to be performed at home at least three times per week, and a walking plan to be undertaken at least two times per week for 24 weeks. . Trained peer mentors will contact and visit the patients at their home to start the exercise programme with them and will follow-up with up to three more home visits / exercise sessions as the participants require
  Arms: OEP
Behavioral: Fame — Community based exercise programme (FaME) FaME includes and extends the OEP. It will comprise one hour PSI delivered group exercise class in a local community centre for a maximum of 15 participants, and two 30 minute home exercise sessions (based on the extended OEP) per week for 24 weeks. Participants will also be advised to walk at least twice per week for up to 30 minutes at a moderate pace.
  Arms: Fame
Other: Treatment As Usual — Treatment as usual by the general practitioner
  Other Names: Usual clinical care
  Arms: TAU

SUMMARY:
The aim of the project is to evaluate the delivery, impact and cost effectiveness of a community based exercise programme (FaME); compared to a home based exercise programme (OEP) supported by similarly aged mentors; compared with usual care for primary care patients.

Primary Objective:

1. To determine the effect on continuation of exercise of two evidence based exercise programmes designed for older people, compared with usual care i.e. with no special interventions to promote physical activity.

   Secondary Objective:
2. To determine the health benefits of the programmes to patients starting at various levels of physical activity, particularly the effects on physical and psychological status, health status and quality adjusted life years (QALYs).
3. To estimate the costs of the exercise interventions and to assess the cost-effectiveness of community group exercise, and home-supported exercise compared with usual care.
4. To determine the acceptability of the programmes, adherence rates, enabling factors and barriers to future implementation.
5. To determine participants' perceptions of the value of exercise, and the predictors of continued exercise.

DETAILED DESCRIPTION:
A cluster controlled trial using minimisation for allocation at the level of general practice in two centres (London and Nottingham/Derby), to compare a community-centre based group exercise programme - FaME [delivered by specifically trained postural stability instructors (PSIs) and supplemented by home exercise and prescriptive recommendations for walking], with a home based exercise programme and walking plan - OEP [supported by specifically trained and similarly aged mentors], with two years follow-up to determine the impact, acceptability and adherence to the programme, and longer term continuation of exercise. Control subjects will continue to receive usual care in primary care. A cost-effectiveness analysis will be conducted within the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be those aged 65+ who can walk around at home (i.e. not chair or bed bound) and would be physically able to take part in a group exercise class, who are not already receiving any long term physiotherapy and who do not fulfill the exclusion criteria.

Exclusion Criteria:

* Chair or bed bound
* Receiving long-term physiotherapy
* Three or more falls in the previous year i.e. frequent fallers (only excluded if their GP does not consent to them taking part in exercise)
* Resting BP > 180/100 mmHg, tachycardia > 100bpm, uncontrolled hypertension
* Significant drop in BP during exercise
* Psychiatric conditions or physical abilities which would prevent participation in an exercise class (for example psychotic illness, acute systemic illness (e.g. pneumonia), uncontrolled visual or vestibular disturbances which the GP considers would exclude patients from undertaking the exercise programme, poorly controlled angina, acute rheumatoid arthritis, unstable or acute heart failure, or conditions requiring a specialist exercise programme e.g. uncontrolled epilepsy significant neurological disease or impairment, unable to maintain seated upright position or unable to move about independently indoors)
* Not living independently (e.g. residential care)
* Significant cognitive impairment (unable to follow simple instructions)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
type, intensity, duration and frequency of physical activity | two years after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Denise Kendrick, PhD, Study Director — University of Nottingham
Locations (2):
- United Kingdom (2):
  - University College London, London
  - University of Nottingham, Nottingham